CLINICAL TRIAL: NCT00818376
Title: Staining And Calculus Formation After 0.12% Chlorhexidine Rinses In Plaque-Free And Plaque-Covered Surfaces. A Randomized Trial.
Brief Title: Staining and Calculus Formation After 0.12% Chlorhexidine Rinses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lutheran University of Brazil (Other)
Responsible Party: Cassiano Kuchenbecker Rösing, Lutheran University Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: LutheranUB
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Dental Calculus; Tooth Discoloration
Keywords: Chlorhexidine; adverse effects; staining; dental calculus; dental plaque
MeSH Terms: conditions — Dental Calculus; Tooth Discoloration; Dental Plaque | interventions — Dental Prophylaxis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Dental prophylaxis — Two randomized quadrants will be cleaned with a prophylaxis to disrupt dental biofilm presence.

SUMMARY:
The presence of plaque on tooth surfaces as a predictor of chlorhexidine side effects has not been evaluated especially because most studies utilized a previous disruption of biofilms in all dental surfaces before the beginning of rinsing. The purpose of this study is to compare staining and calculus formation after 0.12 percent chlorhexidine between previously plaque-free and plaque-covered surfaces by means of an experimental gingivitis model.

DETAILED DESCRIPTION:
Test panel

The test panel will be recruited from the dental students of the Lutheran University of Brazil, Canoas, Rio Grande do Sul, Brazil. At recruitment, subjects will be asked about their medical and dental history. Written and oral explanations detailing the study purpose and design will be given for each subject. Subjects that preliminarily met inclusion/exclusion criteria will be selected for a dental screening appointment. If the subject met all the inclusion/exclusion criteria, an informed consent was handed out and, upon acceptance, signed by the volunteers.

The following clinical parameters were assessed in the order listed below from all teeth, excepting the third higher/lower molar.

Presence of calculus (C) in all teeth, at 6 sites per tooth (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual and disto-lingual) was scored as a dichotomous index: 0 - Absence of calculus; 1 - Presence of calculus.

Discoloration Index proposed by Lobene 36 and modified by Macpherson et al. 2000. This involves visual stain assessment of the buccal/labial and lingual/palatal aspects of the index teeth.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-35 years
* Male
* No relevant medical conditions that could interfere on the periodontal health
* Probing pocket depth < 3 mm and clinical attachment loss < 2mm at all sites
* Willingness to comply

Exclusion Criteria:

* Antibiotic and/or anti-inflammatory therapy within 3 months prior to baseline examination
* Oral mucosal lesions
* Smokers
* Need for antibiotic premedication
* History of hypersensitivity to chlorhexidine
* Any device that could act as plaque retentive factor (e.g., carious lesions, inadequate restorations, dental implants, orthodontic appliances, fixed or removable prostheses)

Exclusion criteria during the study:

* Individuals that wanted to give up the study
* Any acute process like allergic reaction to the product or gingival abcess
* Necessity to use of any antibiotic or anti-inflammatory
* Use of any other rinsing product farther the chlorhexidine's rinses
* Individuals who did any mechanical biofilm control

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-06; Primary Completion 2006-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Dental Staining | 21 days

SECONDARY OUTCOMES:
Dental calculus formation | 21 days

REFERENCES:
- [Derived] Zanatta FB, Antoniazzi RP, Rosing CK. Staining and calculus formation after 0.12% chlorhexidine rinses in plaque-free and plaque covered surfaces: a randomized trial. J Appl Oral Sci. 2010 Sep-Oct;18(5):515-21. doi: 10.1590/s1678-77572010000500015. PMID 21085810